CLINICAL TRIAL: NCT01332435
Title: Dutasteride in Enlarged Prostate Economic Assessment: A Retrospective Database Pooled Analysis of Early 5-alpha Reductase Inhibitor Use
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113984
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2011-07-22 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Prostatic Hyperplasia
Keywords: Enlarged prostate, 5-alpha-reductase inhibitor, alpha-blocker, early, costs
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Early 5ARI Initiation: Patients with EP receiving combination therapy (AB + 5ARI) with early initiation of 5ARI (within 30 days of initiation of AB)
  Interventions: Drug: 5ARI + AB
- Late 5ARI Initiation: Patients with EP receiving combination therapy (AB + 5ARI) with late initiation of 5ARI (more than 30 days but less than 6 months after initiation of AB)
  Interventions: Drug: 5ARI + AB

INTERVENTIONS:
Drug: 5ARI + AB — 5ARI: Dutasteride or Finasteride AB: Doxazosin, Tamsulosin, Terazosin, or Alfuzosin

SUMMARY:
This retrospective study aims to assess the economic impact of early initiation of 5-alpha-reductase inhibitor (5ARI) therapy in patients with enlarged prostate (EP) receiving 5ARI and alpha-blocker (AB) combination therapy. Both the Integrated Health Care Information Solutions and PharMetrics databases will be utilized for this study (2000-2007).

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 50 years or older
* a medical claim of EP
* a prescription claim for a 5ARI and AB (provided both are within 180 days of index date)
* continuously eligible for 6 months prior to and at least 12 months after index prescription date.

Exclusion Criteria:

* diagnosis of prostate or bladder cancer
* any prostate-related surgical procedure within 5 months of index date
* prescription claim for finasteride indicative of male pattern baldness
* 5ARI therapy initiated prior to initiating AB therapy

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to identify eligible patient data between July 1, 2000, and December 31, 2006, and allows for patient data to be followed for 6 months prior to and up to 1 year following index prescription date.
Sampling Method: Probability Sample
Enrollment: 6896 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- IHCIS; Early 5ARI Initiation: Participants from the Integrated Health Care Information Solutions (IHCIS), a nationally representative managed care database that represents over 30 health plans and more than 25 million lives. Early 5ARI Initiation was defined as participants who started on a 5-alpha-reductase inhibitor (5ARI [dutasteride and finasteride]) within 30 days of an alpha-blocker (AB [doxazosin, prazosin, tamsulosin, terazosin, and alfuzosin]).
- IHCIS; Late 5ARI Initiation: Participants from the IHCIS, a nationally representative managed care database that represents over 30 health plans and more than 25 million lives. Late 5ARI Initiation was defined as participants who started on a 5ARI (dutasteride and finasteride) > 30 days after an AB (doxazosin, prazosin, tamsulosin, terazosin, and alfuzosin).
- PharMetrics; Early 5ARI Initiation: Participants from PharMetrics, a database containing data from over 90 different managed healthcare plans, encompassing over 60 million lives. Early 5ARI Initiation was defined as participants who started on a 5ARI (dutasteride and finasteride) within 30 days of an AB (doxazosin, prazosin, tamsulosin, terazosin, and alfuzosin).
- PharMetrics; Late 5ARI Initiation: Participants from PharMetrics, a database containing data from over 90 different managed healthcare plans, encompassing over 60 million lives. Late 5ARI Initiation was defined as participants who started on a 5ARI (dutasteride and finasteride) > 30 days after an AB (doxazosin, prazosin, tamsulosin, terazosin, and alfuzosin).
Period: Overall Study
Arm/Group | IHCIS; Early 5ARI Initiation | IHCIS; Late 5ARI Initiation | PharMetrics; Early 5ARI Initiation | PharMetrics; Late 5ARI Initiation
Started | 1572 | 1064 | 2604 | 1656
Completed | 1572 | 1064 | 2604 | 1656
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IHCIS; Early 5ARI Initiation | IHCIS; Late 5ARI Initiation | PharMetrics; Early 5ARI Initiation | PharMetrics; Late 5ARI Initiation | Total
Number analyzed (Participants) | 1572 | 1064 | 2604 | 1656 | 6896
Age, Customized [Number; unit: Participants]
  >=50 years old | 1572 | 1064 | 2604 | 1656 | 6896
  <50 years old | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 1572 | 1064 | 2604 | 1656 | 6896

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Progression
Description: Clinical progression was identified as the occurrence of acute urinary retention and/or surgery as identified by relevant Common Procedure Terminology (CPT) procedure codes and International Classification of Diseases (ICD)-9CM diagnosis codes.
Time Frame: Day 1 of a 1-day study
Population: Enrolled Population: Men aged >=50 years old between 7/1/2000 and 12/31/2006 with a diagnosis of benign prostatic hyperplasia and who were treated with an AB and concomitant 5-ARI therapy within 6 months of starting AB therapy
Measure: Number; unit: participants
Arm/Group | IHCIS; Early 5ARI Initiation | IHCIS; Late 5ARI Initiation | PharMetrics; Early 5ARI Initiation | PharMetrics; Late 5ARI Initiation
Number analyzed (Participants) | 1572 | 1064 | 2604 | 1656
participants | 176 | 202 | 266 | 232
Statistical Analysis 1: Comparison: IHCIS; Early 5ARI Initiation vs IHCIS; Late 5ARI Initiation; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: PharMetrics; Early 5ARI Initiation vs PharMetrics; Late 5ARI Initiation; Test type: Superiority or Other; p = 0.0002, Chi-squared

2. Primary Outcome: Number of Participants With Acute Urinary Retention
Description: Acute urinary retention was identified by relevant CPT procedure codes and ICD-9CM diagnosis codes.
Time Frame: Day 1 of a 1-day study
Population: Enrolled Population
Measure: Number; unit: participants
Arm/Group | IHCIS; Early 5ARI Initiation | IHCIS; Late 5ARI Initiation | PharMetrics; Early 5ARI Initiation | PharMetrics; Late 5ARI Initiation
Number analyzed (Participants) | 1572 | 1064 | 2604 | 1656
participants | 127 | 140 | 182 | 166
Statistical Analysis 1: Comparison: IHCIS; Early 5ARI Initiation vs IHCIS; Late 5ARI Initiation; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: PharMetrics; Early 5ARI Initiation vs PharMetrics; Late 5ARI Initiation; Test type: Superiority or Other; p = 0.0006, Chi-squared

3. Primary Outcome: Number of Participants Who Needed Prostate-Related Surgery
Description: Prostate-related surgery was identified by relevant CPT procedure codes and ICD-9CM diagnosis codes.
Time Frame: Day 1 of a 1-day study
Population: Enrolled Population
Measure: Number; unit: participants
Arm/Group | IHCIS; Early 5ARI Initiation | IHCIS; Late 5ARI Initiation | PharMetrics; Early 5ARI Initiation | PharMetrics; Late 5ARI Initiation
Number analyzed (Participants) | 1572 | 1064 | 2604 | 1656
participants | 75 | 101 | 130 | 104
Statistical Analysis 1: Comparison: IHCIS; Early 5ARI Initiation vs IHCIS; Late 5ARI Initiation; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: PharMetrics; Early 5ARI Initiation vs PharMetrics; Late 5ARI Initiation; Test type: Superiority or Other; p = 0.0699, Chi-squared

4. Secondary Outcome: Total BPH-related Costs
Description: All costs related to BPH were defined by claims costs associated with a ICD-9CM diagnosis code for BPH (222.2, 600.xx).
Time Frame: Day 1 of a 1-day study
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | IHCIS; Early 5ARI Initiation | IHCIS; Late 5ARI Initiation | PharMetrics; Early 5ARI Initiation | PharMetrics; Late 5ARI Initiation
Number analyzed (Participants) | 1572 | 1064 | 2604 | 1656
United States dollars | 1417 (1670) | 1606 (1878) | 1735 (1687) | 1686 (2098)
Statistical Analysis 1: Comparison: IHCIS; Early 5ARI Initiation vs IHCIS; Late 5ARI Initiation; Test type: Superiority or Other; p < 0.001, Regression, Linear
Statistical Analysis 2: Comparison: PharMetrics; Early 5ARI Initiation vs PharMetrics; Late 5ARI Initiation; Test type: Superiority or Other; p = 0.8645, Regression, Linear

5. Secondary Outcome: BPH-related Medical Costs
Description: Medical costs related to BPH were defined by claims costs associated with a ICD-9CM diagnosis code for BPH (222.2, 600.xx).
Time Frame: Day 1 of a 1-day study
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | IHCIS; Early 5ARI Initiation | IHCIS; Late 5ARI Initiation | PharMetrics; Early 5ARI Initiation | PharMetrics; Late 5ARI Initiation
Number analyzed (Participants) | 1572 | 1064 | 2604 | 1656
United States dollars | 349 (1535) | 618 (1812) | 344 (1458) | 449 (2001)
Statistical Analysis 1: Comparison: IHCIS; Early 5ARI Initiation vs IHCIS; Late 5ARI Initiation; Test type: Superiority or Other; p < 0.001, Regression, Linear
Statistical Analysis 2: Comparison: PharMetrics; Early 5ARI Initiation vs PharMetrics; Late 5ARI Initiation; Test type: Superiority or Other; p < 0.001, Regression, Linear

6. Secondary Outcome: BPH-related Pharmacy Costs
Description: Pharmacy costs related to BPH were defined by claims costs associated with a ICD-9CM diagnosis code for BPH (222.2, 600.xx).
Time Frame: Day 1 of a 1-day study
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | IHCIS; Early 5ARI Initiation | IHCIS; Late 5ARI Initiation | PharMetrics; Early 5ARI Initiation | PharMetrics; Late 5ARI Initiation
Number analyzed (Participants) | 1572 | 1064 | 2604 | 1656
United States dollars | 1068 (645) | 1417 (1670) | 1392 (851) | 1237 (733)

ADVERSE EVENTS:
Description: This was a retrospective database study, and adverse event/serious adverse event information was not captured in the study.
Arm/Group | IHCIS; Early 5ARI Initiation | IHCIS; Late 5ARI Initiation | PharMetrics; Early 5ARI Initiation | PharMetrics; Late 5ARI Initiation
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.